CLINICAL TRIAL: NCT03465956
Title: Laparoscopic Sleeve Gastrectomy Short Term Follow up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Gamal Thabet (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Gamal Thabet, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed gamal
Record Dates: First submitted 2018-02-21; First posted 2018-03-15 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: All patients,males and females with age (20-50 years old) with morbid obesity (BMI ≥ 40 kg/m2 or > 35 kg/m2 associated with co-morbidity).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Sleeve Gastrectomy (Other): Laparoscopic sleeve gastrectomy for patients with morbid obesity using the gastro-intestinal anastomosis stapler.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy using the gastro-intestinal anastomosis stapler.

SUMMARY:
Laparoscopic Sleeve Gastrectomy (LSG), Also known as longitudinal or vertical gastrectomy.

LSG was initially considered a first-stage operation in high-risk patients before bilio-pancreatic diversion or Roux-en-Y gastric bypass surgery. However, LSG was subsequently found to be effective as a single procedure for treatment of morbid obesity.LSG functions mainly as a restrictive procedure in which about 75 % of the stomach is removed leaving a narrow gastric tube or sleeve. So, it limits the amount of food that can be eaten at one time via inducing early satiety after eating a small amount of food due to early distension of the fashioned gastric sleeve giving a sense of satiety, consequently losing excess body weight by time.Sleeve gastrectomy may also cause a decrease in appetite by reducing the amount of Ghrelin (hunger hormone) produced by the stomach.

DETAILED DESCRIPTION:
All patients,males and females with age (20-50 years old) with morbid obesity (BMI ≥ 40 kg/m2 or > 35 kg/m2 associated with co-morbidity) randomly admitted to Assiut University Hospital-General Surgery Department.

Pre-operative: Assessment of; BMI (Body Mass Index), Fasting Blood Glucose level (FBG), Associated Co-morbidities (as hypertensions & sleep apnea).

Operative (During Operation):

All patients undergo LSG by single team work with intra-operative oesophageal bougie 36 french with use of laparoscopic gastro-intestinal anastomosis(GIA) stapler.

Post-operative:

Patients are discharged from the hospital after they can start oral diet.

Post-operative evaluation of:

1. Complications:

   1. Early complications: during the first 2 weeks after surgery,which include hemorrhage (intra-luminal or extra-luminal), staple line leak, vomiting and infection (surgical site infection or intra- abdominal abscess formation)
   2. Late complications: from 2 weeks to 6 months post-operative, which include stricture of the gastric sleeve, gastro-esophageal reflux disease (GERD) and nutritional deficiencies.
2. Excess weight loss (EWL) by using BMI Follow up of patients at fifteen days, one month, two months, three months and six months after surgery.
3. Assessment of Blood Glucose level during visits.
4. Measurement of blood pressure during visits (if there is associated hypertension).

ELIGIBILITY:
Inclusion Criteria:

* All patients,males and females with age (20-50 years old) with morbid obesity (BMI ≥ 40 kg/m2 or > 35 kg/m2 associated with co-morbidity), and are fit for laparoscopic surgery.

Exclusion Criteria:

* Patients having severe co-morbidity who are not fit for surgery or general anaesthesia.
* Patients with age below 20 years or above 50 years.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of excess weight loss | First six months after surgery
  Assessment of excess weight loss six months after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gamal, Principal Investigator — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nosso G, Angrisani L, Saldalamacchia G, Cutolo PP, Cotugno M, Lupoli R, Vitolo G, Capaldo B. Impact of sleeve gastrectomy on weight loss, glucose homeostasis, and comorbidities in severely obese type 2 diabetic subjects. J Obes. 2011;2011:340867. doi: 10.1155/2011/340867. Epub 2011 Mar 8. PMID 21423553